CLINICAL TRIAL: NCT05724199
Title: A Phase 3, Randomized, 24-week, Placebo-controlled, Double-blind Study to Assess the Efficacy, Safety, and Tolerability of Rocatinlimab (AMG 451) in Combination With Topical Corticosteroids and/or Topical Calcineurin Inhibitors in Adult Subjects With Moderate-to-severe Atopic Dermatitis (AD) (ROCKET-SHUTTLE)
Brief Title: A Study Assessing Rocatinlimab in Combination With Topical Corticosteroid and/or Topical Calcineurin Inhibitors in Adult Participants With Moderate-to-severe Atopic Dermatitis (AD)
Acronym: ROCKET-SHUTTLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20210144; 2022-501585-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; AMG 451; Eczema; Rocatinlimab; KHK4083
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Rocatinlimab Dose 1 + TCS/TCI (Experimental): Rocatinlimab Dose 1 every 4 weeks (Q4W) for 24 weeks + TCS/TCI + loading dose at Week 2.
  Interventions: Drug: Rocatinlimab
- Rocatinlimab Dose 2 + TCS/TCI (Experimental): Rocatinlimab Dose 2 Q4W for 24 weeks + TCS/TCI + loading dose at Week 2.
  Interventions: Drug: Rocatinlimab
- Placebo + TCS/TCI (Placebo Comparator): Placebo Q4W for 24 weeks + TCS/TCI + loading dose at Week 2.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rocatinlimab — Subcutaneous (SC) injection
  Other Names: AMG 451
  Arms: Rocatinlimab Dose 1 + TCS/TCI; Rocatinlimab Dose 2 + TCS/TCI
Other: Placebo — SC injection
  Arms: Placebo + TCS/TCI

SUMMARY:
The coprimary objectives of the study are to:

* evaluate the efficacy of rocatinlimab in combination with topical corticosteroid and/or topical calcineurin inhibitor (TCS/TCI), compared with placebo in combination with TCS/TCI at Week 24, assessed using Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD™).
* evaluate the efficacy of rocatinlimab, in combination with TCS/TCI, compared with placebo in combination with TCS/TCI at Week 24, assessed using Eczema Area and Severity Index (EASI).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with a diagnosis of AD according to the AAD (American Academy of Dermatology) Consensus Criteria (2014) present for at least 12 months
* History of inadequate response to TCS of medium or higher potency (with or without TCI)
* EASI score ≥16
* vIGA-AD score ≥3
* ≥10% body surface area (BSA) of AD involvement
* Worst pruritus numerical rating scale ≥ 4

Exclusion Criteria:

* Treatment with a biological product within 12 weeks or 5 half-lives, whichever is longer, prior to Day 1
* Treatment with any of the following medications or therapies within 4 weeks or 5 half-lives, whichever is longer, prior to Day 1:

  * Systemic corticosteroids
  * Nonbiologic, non-targeted Systemic immunosuppressants
  * Phototherapy
  * Janus kinase inhibitors
* Treatment with any of the following medications or therapies within 1 week, prior to Day 1:

  * TCS
  * TCI
  * Topical phosphodiesterase type 4 inhibitors
  * Other topical immunosuppressive agents
  * Combination topical agents including TCS of any potency or TCI, PDE4 inhibitors, or other topical immunosuppressive agents

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Achievement of a vIGA-AD Score of 0 or 1 with a ≥2 Point Reduction From Baseline at Week 24 | Baseline, Week 24
Achievement of ≥ 75% Reduction From Baseline in EASI Score (EASI 75) at Week 24 | Baseline, Week 24

SECONDARY OUTCOMES:
Achievement of EASI 75 at Week 16 | Baseline, Week 16
Achievement of vIGA-AD 0/1 at Week 16 | Baseline, Week 16
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of Daily Worst Pruritus Numeric Rating Scale (NRS) Score at Week 16 in Participants with Baseline Weekly Average of Daily Worst Pruritus NRS Score ≥ 4 | Baseline, Week 16
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 24 in Participants with Baseline Weekly Average of Daily Worst Pruritus NRS Score ≥ 4 | Baseline, Week 24
Achievement of ≥ 90% Reduction From Baseline in EASI Score (EASI 90) at Week 24 | Baseline, Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of AD Skin Pain NRS Score at Week 24 in Participants With Baseline Weekly Average of AD Skin Pain NRS Score ≥ 4 | Baseline, Week 24
Achievement of vIGA-AD 1 Response with a Presence of Only Barely Perceptible Erythema or vlGA-AD 0 Response (Revised IGA [rIGA™] 0/1) at Week 24 | Baseline, Week 24
Achievement of a Facial AD Severity Score of Clear at Week 24 for Participants with Facial AD at Baseline | Baseline, Week 24
Achievement of a Hand AD Severity Score of Clear at Week 24 for Participants with Hand AD at Baseline | Baseline, Week 24
Change From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 16 | Baseline, Week 16
Change From Baseline in Weekly Average of Daily Worst Pruritus NRS Score at Week 24 | Baseline, Week 24
Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Itch Visual Analogue Scale (VAS) Score at Week 16 | Baseline, Week 16
Change From Baseline in SCORAD Itch VAS Score at Week 24 | Baseline, Week 24
Achievement of ≥ 4-point Reduction From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 24 in Participants With Baseline DLQI Score ≥ 4 | Baseline, Week 24
Change from Baseline in DLQI Score at Week 24 | Baseline, Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Patient Oriented Eczema Measure (POEM) Score at Week 24 in Participants with Baseline POEM Score ≥ 4 | Baseline, Week 24
Change From Baseline in POEM Score at Week 24 | Baseline, Week 24
Achievement of a ≥ 4-point Reduction From Baseline in Weekly Average of AD Skin Pain NRS Score at Week 16 in Participants With Baseline Weekly Average of AD skin pain NRS Score ≥ 4 | Baseline, Week 16
Change From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 24 | Baseline, Week 24
Change From Baseline in Weekly Average of Daily AD Skin Pain NRS Score at Week 16 | Baseline, Week 16
Achievement of a ≥ 3-point Reduction From Baseline in Weekly Average of AD Skin Pain NRS Score at Week 24 in Participants With Baseline Weekly Average of AD Skin Pain NRS Score ≥ 3 | Baseline, Week 24
Achievement of a ≥ 3-point Reduction From Baseline in Weekly Average of AD Skin Pain NRS Score at Week 16 in Participants With Baseline Weekly Average of AD Skin Pain NRS Score ≥ 3 | Baseline, Week 16
Change From Baseline in Weekly Average of Sleep Disturbance NRS Score at Week 24 | Baseline, Week 24
Achievement of a Hospital Anxiety and Depression Scale (HADS)-anxiety Subscale Score < 8 at Week 24 in Participants with Baseline HADS-anxiety Subscale Score ≥ 8 | Baseline, Week 24
Achievement of a HADS-depression Subscale Score < 8 at Week 24 in Participants with Baseline HADS-depression Subscale Score ≥ 8 | Baseline, Week 24
Change From Baseline in HADS-anxiety Subscale Score at Week 24 | Baseline, Week 24
Change From Baseline in HADS-depression Subscale Score at Week 24 | Baseline, Week 24
Achievement of a ≥ 8.7-point Reduction from Baseline in SCORAD Score at Week 24 in Participants with Baseline SCORAD Score ≥ 8.7 | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (234):
- United States (45):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Medical Dermatology Specialists, Phoenix, Arizona
  - Southwest Skin Specialists, Phoenix, Arizona
  - US Dermatology Partners Sun City West, Sun City West, Arizona
  - Arkansas Research Trials, LLC, North Little Rock, Arkansas
  - Kern Research Inc, Bakersfield, California
  - Keck Medicine of University of Southern California, Los Angeles, California
  - Wallace Medical Group Inc, Los Angeles, California
  - Antelope Valley Clinical Trials, Palmdale, California
  - University of California at Davis Medical Center, Sacramento, California
  - Kaiser Permanente South Sacramento Medical Center, Sacramento, California
  - Acclaim Clinical Research, San Diego, California
  - Kaiser Permanente Medical Center - Oakland, San Francisco, California
  - Kaiser Permanente Medical Center - San Francisco, San Francisco, California
  - Synergy Dermatology, San Francisco, California
  - TrueBlue Clinical Research, Tampa, Florida
  - Olympian Clinical Research - Tampa, Tampa, Florida
  - Atlanta Dermatology, Vein and Research Center, PC, Alpharetta, Georgia
  - Divine Dermatology and Aesthetics, Atlanta, Georgia
  - NorthShore University HealthSystem, Skokie, Illinois
  - DS Research, Clarksville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dermatology and Skin Cancer Center Leawood, Leawood, Kansas
  - Industrial Medicine Associates Clinical Research Advanced Dermatology Care, Monroe, Louisiana
  - Aesthetic and Dermatology Center, Rockville, Maryland
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - Somnos Clinical Research, Lincoln, Nebraska
  - Skin Specialists PC, Omaha, Nebraska
  - Vivida Dermatology, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Schweiger Dermatology Group, PC Research Division, Hackensack, New Jersey
  - Albuquerque Clinical Trials Incorporated, Albuquerque, New Mexico
  - Chear Center LLC, The Bronx, New York
  - Accellacare of Wilmington, Wilmington, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Velocity Clinical Research Inc, Medford, Oregon
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - US Dermatology Partners Jollyville, Austin, Texas
  - Newco 3A Research LLC, El Paso, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Texas Dermatology Research Center, Plano, Texas
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
- Argentina (8):
  - Cinme - Centro de Investigaciones Metabolicas, CABA, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - Dim Clinica Privada, Ramos Mejía, Buenos Aires
  - Buenos Aires Skin SA, Buenos Aires, Distrito Federal
  - Fundacion Cidea, Buenos Aires, Distrito Federal
  - Care- Centro de Alergia y Enfermedades Respiratorias, Buenos Aires, Distrito Federal
  - Psoriahue Medicina Interdisciplinaria SRL, Buenos Aires, Distrito Federal
  - Centro de Investigaciones Clinicas Instituto Especialidades De La Salud De Rosario, Rosario, Santa Fe Province
- Australia (6):
  - Emeritus Research Sydney, Botany, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Princess Alexandra Hospital, South Brisbane, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Emeritus Research Melbourne, Camberwell, Victoria
- Austria (5):
  - Medizinische Universitaet Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Landeskrankenhaus Salzburg, Salzburg
  - Klinik Landstrasse, Vienna
  - Klinik Hietzing, Vienna
- Belgium (10):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende, Bruges
  - Centre Hospitalier Universitaire Brugmann, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universite Catholique de Louvain Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Clinique Andre Renard, Herstal
  - Dermatologie Handelskaai, Kortrijk
  - Universitaire Ziekenhuizen Leuven Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Grand Hopital de Charleroi, Loverval
- Bulgaria (5):
  - Medical Center Asklepii OOD, Dupnitsa
  - Medical Center Medconsult Pleven OOD, Pleven
  - Medical Center Excelsior OOD, Sofia
  - Diagnostic-Consultative Center Alexandrovska EOOD, Sofia
  - Diagnostic-Consultative Center - Fokus-5 - Medical Institution for Outpatient Care OOD, Sofia
- Canada (21):
  - Dermatology Research Institute Incorporated, Calgary, Alberta
  - Laser Rejuvenation Clinics Edmonton D T Incorporated, Edmonton, Alberta
  - Alberta Derma Surgery Centre, Edmonton, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Incorporated, Winnipeg, Manitoba
  - SKiN Health, Coburg, Ontario
  - Centricity Research London, London, Ontario
  - Dr SK Siddha Medicine Professional Corporation, Newmarket, Ontario
  - Allergy Research Canada Incorporated, Niagara Falls, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - JRB Research Incorporated, Ottawa, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - North York Research Incorporated, Toronto, Ontario
  - Toronto Research Centre Inc, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - Clinique de Dermatologie Rosemont, Montreal, Quebec
  - Innovaderm Research Inc, Montreal, Quebec
  - DIEX Recherche Quebec, Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec, Quebec
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan
- China (21):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital ,Sun-Yat Sen University, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The Fist Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Qianhai Shekou Free Trade Zone Hospital, Shenzhen, Guangdong
  - Nanyang First Peoples Hospital, Nanyang, Henan
  - Union Hospital Tongji Medical College Huazhong University of science and Technology, Wuhan, Hubei
  - Wuxi Second Peoples Hospital, Wuxi, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
  - the First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Affiliated Hangzhou First Peoples Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliation Hospital Of Ningbo University, Ningbo, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - Peking University Peoples Hospital, Beijing
  - Shanghai Skin Disease Hospital, Shanghai
- France (17):
  - Hopital Prive d Antony, Antony
  - Centre Hospitalier Universitaire de Bordeaux - Hôpital Saint André, Bordeaux
  - Centre Hospitalier Regional Universitaire Brest Hopital Morvan, Brest
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille
  - Centre Hospitalier de Bretagne Sud - Hopital du Scorff, Lorient
  - Hôpital La Timone, Marseille
  - Cabinet du Docteur Ruer-Mulard Mireille, Martigues
  - Centre Hospitalier Universitaire de Nantes Hôtel Dieu, Nantes
  - Centre Hospitalier Universitaire Archet 2, Nice
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Tenon, Paris
  - Hopital Saint Louis, Paris
  - Polyclinique de Courlancy, Reims
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Rouen - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - Hopital d instruction des armees sainte anne, Toulon
- Germany (10):
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Universitaetsmedizin Goettingen - Georg-August-Universitaet, Göttingen
  - TFS Trial Form Support GmbH, Hamburg
  - MensingDerma research GmbH, Hamburg
  - Hautaerzte Zentrum Hannover, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsmedizin Mainz, Mainz
  - Beldio Research GmbH, Memmingen
  - Hautmedizin Saar, Merzing
  - Klinikum rechts der Isar der TUM, München
- Greece (6):
  - 401 General Military Hospital Of Athens, Athens
  - Andreas Syngros Hospital Of Venereal And Dermatological Diseases, Athens
  - University General Hospital of Heraklion, Heraklion
  - General Hospital Of Nea Ionia Konstantopouleio Patision, Nea Ionia
  - Geniko Nosokomeio Peiraia Tzaneio, Piraeus
  - Ippokratio General Hospital of Thessaloniki, Thessaloniki
- Hungary (10):
  - Trial Pharma Kft, Békéscsaba
  - Csalogany Orvosi Kozpont, Budapest
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz, Kaposvár
  - DermaMed Research Kft, Orosháza
  - Allergo-Derm Bakos Kft, Szolnok
  - Obudai Egeszsegugyi Centrum Kft, Zalaegerszeg
- Italy (4):
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Ospedale San Salvatore, LAquila
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano MI
- Japan (15):
  - Fukui Dermatology Clinic, Nagoya, Aichi-ken
  - Ekihigashi Dermatology Allergy Clinic, Fukuoka, Fukuoka
  - Takagi Dermatological Clinic Branch, Obihiro-shi, Hokkaido
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hokkaido
  - Katahira Dermatology Urology Clinic, Kagoshima, Kagoshima-ken
  - Kosugi Dermatology Clinic, Kawasaki-shi, Kanagawa
  - Nomura Dermatology Clinic, Yokohama, Kanagawa
  - Jouzan Hihuka Hinyoukika Clinic, Kumamoto, Kumamoto
  - Suizenji Dermatology Clinic, Kumamoto, Kumamoto
  - Yoshioka Dermatology Clinic, Neyagawa, Osaka
  - JA Shizuoka Kohseiren Enshu Hospital, Hamamatsu, Shizuoka
  - Mildix Skin Clinic, Adachi-ku, Tokyo
  - Naoko Dermatology Clinic, Setagaya-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Yamate Dermatology Clinic, Shinjuku-ku, Tokyo
- Malaysia (7):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
- Netherlands (3):
  - Bravis Ziekenhuis, Bergen op Zoom
  - Universitair Medisch Centrum Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (7):
  - Dermapolis Medical Dermatology Center dr n med Edyta Gebska, Chorzów
  - GynCentrum Spzoo NZOZ Holsamed - Oddzial Libero, Katowice
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno-Badawczy Marek Brzewski Pawel Brzewski SpCywilna, Krakow
  - AppleTreeClinics Network Spzoo, Lodz
  - Ip Clinic Sp zoo, Lodz
  - Twoja Przychodnia Scm, Szczecin
  - DermMedica Spzoo Centrum Columbus, Wroclaw
- Doctor Samuel Sanchez PSC, Caguas, Puerto Rico
- Romania (3):
  - Theramed Healthcare SRL, Brasov
  - Institutul Regional de Gastroenterologie si Hepatologie Prof Dr Octavian Fodor, Cluj-Napoca
  - Spitalul Clinic Judetean Mures, Târgu Mureş
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Skin Centre, Singapore
- Slovakia (4):
  - Maxderm, sro, Bardejov
  - Univerzitna nemocnica Bratislava - Nemocnica Stare Mesto, Bratislava
  - Fakultna nemocnica s poliklinikou JA Reimana Presov, Prešov
  - Sanare spol sro, Svidník
- Slovenia (2):
  - Univerzitetni klinicni center Ljubljana, Ljubljana
  - Univerzitetni Klinicni Center Maribor, Maribor
- Spain (5):
  - Hospital Universitario Basurto, Bilbao, Basque Country
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario 12 de Octubre, Madrid
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
- Switzerland (5):
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Universitaetsspital Zuerich, Zurich
- Turkey (Türkiye) (5):
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Acibadem Altunizade Hastanesi, Istanbul
  - Marmara Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (6):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Russells Hall Hospital, Dudley
  - West Middlesex University Hospital, Isleworth
  - The Royal Free Hospital, London
  - Salford Care Organisation, Salford
  - Accellacare Yorkshire, Shipley

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1)the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Guttman-Yassky E, Simpson E, Bissonnette R, Eichenfield LF, Kabashima K, Luna PC, Hercogova JT, Spelman L, Worm M, Esfandiari E, Arai T, Mano H, Charuworn P, Wang A, Kricorian G. ROCKET: a phase 3 program evaluating the efficacy and safety of rocatinlimab in moderate-to-severe atopic dermatitis. Immunotherapy. 2025 Feb;17(2):83-94. doi: 10.1080/1750743X.2025.2464528. Epub 2025 Feb 26. PMID 40012373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com